CLINICAL TRIAL: NCT02788955
Title: Decreasing the Burden of Sarcopenia in Cancer Through Targeted Nutrition Intervention: A Feasibility Study
Brief Title: Protein Recommendation to Increase Muscle
Acronym: PRIMe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canada Foundation for Innovation (Other); Government of Alberta (Other Government); Nestlé Health Science Spain (Industry); Olymel (Unknown); Cargill (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREBA.CC-15-0193
Record Dates: First submitted 2016-03-23; First posted 2016-06-02 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer
Keywords: Protein; Diet intervention; Muscle; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Dietary Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Protein Diet (Active Comparator): In the normal protein diet, participants will be instructed to follow a diet that will provide them with the amount of calories enough to meet their energy needs without changing their body weight and will contain 1 g of protein per kilogram of body weight. Participants will be instructed to consume protein primarily from animal food sources. A high quality whey protein supplement will be provided as needed.
  Interventions: Behavioral: Dietary counselling; Other: Dietary Protein
- High Protein Diet (Experimental): In the high protein diet, participants will be instructed to follow a diet that will provide them with the amount of calories enough to meet their energy needs without changing their body weight and will contain 2 g of protein per kilogram of body weight. Participants will be instructed to consume protein primarily from animal food sources. A high quality whey protein supplement will be provided as needed.
  Interventions: Behavioral: Dietary counselling; Other: Dietary Protein

INTERVENTIONS:
Behavioral: Dietary counselling
Other: Dietary Protein

SUMMARY:
This is a feasibility study to test the potential efficacy of diets of different amounts of protein and calories for patients with cancer. We hypothesize that nutritional deficits play a significant role in muscle loss and that nutritional therapy is an important first step in reversing or preventing muscle loss and maintaining/improving physical function.

DETAILED DESCRIPTION:
Severe muscle depletion (sarcopenia) is a common issue among cancer patients and adequate nutrient intake is pivotal to maintain muscle mass. Yet, optimal amounts of protein are undefined for preventing or treating sarcopenia in people with cancer as most methodological approaches to assess protein requirements are expensive, burdensome and unfeasible for this population. This study's overarching goal is to investigate the potential efficacy of diets of different protein content on: 1) muscle mass maintenance (primary endpoint); and 2) improvements on physical function in cancer patients capable of oral nutrition support. Additional study measurements include: energy metabolism (including total body), body composition using multi-compartment models, blood biomarkers, and quality of life.

In a randomized controlled trial approach, we will employ high protein feeding (2 g/kg/d, n=16) versus a standard recommendation (1 g/kg/d, n=16) in patients with newly diagnosed colorectal cancer for 12 weeks. Prescribed energy intakes will be framed by the amount of calories to meet energy needs and to support protein synthesis, but prevent fat mass gain. Carbohydrate, fat and protein intake will be adjusted throughout the intervention to achieve the desired rate and amount of energy and protein intake. An oral protein powder supplement made from high-quality whey protein will be provided to the participants to help increase their protein intake as needed. A multivitamin will be given to all participants throughout the study. Participants will receive weekly calls from the study coordinator to ensure adherence to the dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adults 18 - 85 years of age;
* Able to communicate in English;
* Recent diagnosis of colorectal cancer (stage II, III or IV);
* Able to complete all baseline assessments within 2 weeks of commencement of chemotherapy or chemoradiotherapy (when applicable);
* ≥1 year life expectancy and believed to be able to complete 12 weeks of intervention (based on clinical judgment);
* Able to provide a blood sample;
* Adequate hepatic function, as confirmed by medical records and to be checked with patient's oncologist;
* Adequate renal function, as confirmed by medical records and to be checked with patient's oncologist;
* If a woman of childbearing potential, she must agree to use an effective form of contraception during the study (are considered effective forms of contraception: abstinence, a hormonal contraceptive, or a double-barrier method).

Exclusion Criteria:

* Acute inflammation assessed by neutrophil/leukocyte ratio or in consultation with oncologist;
* Ongoing (non-treatment related) nutritional impact symptoms that would impact ability to follow dietary recommendations (ie. anorexia);
* Severe food restrictions (severe food allergy or dietary pattern - e.g. vegetarian);
* Current medical condition that impacts the patients ability to take part in study or impacts the ability to increase muscle (e.g. cachexia, post-surgical wound infection, muscular dystrophy or any degenerative muscle disease or condition);
* Individuals with pacemakers;
* Comorbidities: active treatment for another cancer site, major chronic conditions that would interfere with dietary restriction such as recent myocardial infarction, unstable angina, stroke, or unstable disease such as congestive heart failure;
* Women who are pregnant or breast-feeding;
* Body weight > 450 lb due to limit of body composition measurement instrumentation;
* Presenting with any health condition that would severely affect nutrient absorption (e.g.: enteric fistula);
* Patients diagnosed with metabolic disorders in consultation with the oncologist (e.g. uncontrolled diabetes, recent diagnosis (< 3 months) thyroid disease);
* Cognitive impairment or dementia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Change/maintenance in muscle mass | Baseline, week 12
  To assess the change in muscle mass from baseline to week 12 using Dual-energy X-ray absorptiometry (DXA).

SECONDARY OUTCOMES:
Change in physical function | Baseline, week 12
  To assess the change in total score on the Short Performance Physical Battery (SPPB) test from baseline to week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Prado, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Cross Cancer Institute, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prado CM, Lieffers JR, McCargar LJ, Reiman T, Sawyer MB, Martin L, Baracos VE. Prevalence and clinical implications of sarcopenic obesity in patients with solid tumours of the respiratory and gastrointestinal tracts: a population-based study. Lancet Oncol. 2008 Jul;9(7):629-35. doi: 10.1016/S1470-2045(08)70153-0. Epub 2008 Jun 6. PMID 18539529
- [Background] Prado CM, Lieffers JR, Bowthorpe L, Baracos VE, Mourtzakis M, McCargar LJ. Sarcopenia and physical function in overweight patients with advanced cancer. Can J Diet Pract Res. 2013 Summer;74(2):69-74. doi: 10.3148/74.2.2013.69. PMID 23750978
- [Background] Prado CM, Lieffers JR, Bergsten G, Mourtzakis M, Baracos VE, Reiman T, Sawyer MB, McCargar LJ. Dietary patterns of patients with advanced lung or colorectal cancer. Can J Diet Pract Res. 2012 Winter;73(4):e298-303. doi: 10.3148/73.4.2012.e298. PMID 23217447
- [Background] Prado CM, Cushen SJ, Orsso CE, Ryan AM. Sarcopenia and cachexia in the era of obesity: clinical and nutritional impact. Proc Nutr Soc. 2016 May;75(2):188-98. doi: 10.1017/S0029665115004279. Epub 2016 Jan 8. PMID 26743210
- [Background] Ford KL, Arends J, Atherton PJ, Engelen MPKJ, Goncalves TJM, Laviano A, Lobo DN, Phillips SM, Ravasco P, Deutz NEP, Prado CM. The importance of protein sources to support muscle anabolism in cancer: An expert group opinion. Clin Nutr. 2022 Jan;41(1):192-201. doi: 10.1016/j.clnu.2021.11.032. Epub 2021 Nov 29. PMID 34891022
- [Background] Ford KL, Sawyer MB, Trottier CF, Ghosh S, Deutz NEP, Siervo M, Porter Starr KN, Bales CW, Disi IR, Prado CM. Protein Recommendation to Increase Muscle (PRIMe): Study protocol for a randomized controlled pilot trial investigating the feasibility of a high protein diet to halt loss of muscle mass in patients with colorectal cancer. Clin Nutr ESPEN. 2021 Feb;41:175-185. doi: 10.1016/j.clnesp.2020.11.016. Epub 2020 Dec 24. PMID 33487262
- [Derived] Ford KL, Quintanilha M, Trottier CF, Wismer W, Sawyer MB, Siervo M, Deutz NEP, Vallianatos H, Prado CM. Exploring relationships with food after dietary intervention in patients with colorectal cancer: a qualitative analysis from the Protein Recommendations to Increase Muscle (PRIMe) trial. Support Care Cancer. 2024 Jun 7;32(7):418. doi: 10.1007/s00520-024-08620-1. PMID 38849604
- [Derived] Ford KL, Pichard C, Sawyer MB, Trottier CF, Disi IR, Purcell SA, Ghosh S, Siervo M, Deutz NE, Prado CM. Total energy expenditure assessed by 24-h whole-room indirect calorimeter in patients with colorectal cancer: baseline findings from the PRIMe study. Am J Clin Nutr. 2023 Aug;118(2):422-432. doi: 10.1016/j.ajcnut.2023.06.002. Epub 2023 Jun 7. PMID 37290740